CLINICAL TRIAL: NCT07120373
Title: An Exploration of the Relationship Between Sleep Disturbance, Mental Health, and Functional Outcomes in Mild, Moderate and Severe Traumatic Brain Injury (TBI): A Mixed Methods Study
Brief Title: An Exploration of Sleep Disturbance and Outcomes in TBI (SLEEP-TBI)
Acronym: SLEEP-TBI
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nottingham (Other)
Collaborators: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 25028; 357334 (Other: IRAS Project ID)
Record Dates: First submitted 2025-07-03; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-06

CONDITIONS: Traumatic Brain Injury
Keywords: Sleep disturbance; Head injury; Traumatic brain injury; Sleep; Actigraphy; TBI
MeSH Terms: conditions — Brain Injuries, Traumatic; Parasomnias; Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Part 1: Part 1 - Early Sleep Study - Cohort Study 'Part 1' will consist of a cohort study, in which participants are recruited from Nottingham University Hospitals Trust, within 12 weeks of sustaining their injury. The purpose of this study will be to understand the relationship between early sleep disturbance and recovery in TBI, including understanding the impact on functional recovery and mental health at 3- and 6-months post-injury.
  A combination of subjective data (e.g. sleep diaries and questionnaires) and objective data (actigraphy to measure sleep disturbance via the GENEActiv wrist-worn device) will be used to measure recovery from TBI and sleep disturbance.
- Part 2: Part 2 - Chronic Sleep Study - Cross-sectional 'Part 2' will consist of a cross-sectional study, in which participants are recruited from Nottingham University Hospitals Trust rehabilitation teams, at over 12 months after sustaining their TBI. The purpose of this study will be to understand the relationship between chronic sleep disturbance and recovery in TBI, including functional recovery and mental health. Within this study, we will also consider how these factors may impact on engagement with rehabilitation, as rated by a clinician. A combination of subjective data (e.g. sleep diaries and questionnaires) and objective data (actigraphy to measure sleep disturbance via the GENEActiv wrist-worn device) will be used to measure recovery from TBI and sleep disturbance.
- Part 3: Part 3 - Interviews 'Part 3' will consist of semi-structured interviews with a sub-sample of participants from Parts 1 and 2. The purpose of this study will be to understand and explore the human experience of sleep disturbance and recovery in TBI.

SUMMARY:
This study aims to look at how sleep disturbance affects people who have had a traumatic brain injury.

Sleep disturbance can include waking frequently in the night, difficulty falling asleep, excessive sleepiness or changes to usual sleep patterns.

Investigators define traumatic brain injury as an injury caused by a forceful bump, blow, or jolt to the head or body, or from an object entering the brain. This results in a disturbance of normal brain function, that can be temporary.

By understanding the relationship between sleep disturbance and traumatic brain injury, investigators will hopefully improve care and treatment for people with a traumatic brain injury.

Investigators are looking to understand each participant's experience of sleep disturbance, as well as measuring sleep, using a device that monitors movement and sleep quality.

Investigators are interested how sleep disturbance impacts things like day-to-day life and activities, such as work or leisure. Investigators are also interested in mental health, such as depression or anxiety.

DETAILED DESCRIPTION:
The focus of the study will be to determine whether sleep data acquired longitudinally over the months following traumatic brain injury (TBI) predicts long-term mental health and functional outcomes, including return to normal activities, such as work. The overarching aim is to improve the care and treatment that people with TBI experience, by understanding the predictive value of sleep disturbances.

Overall research aim

The overall aim of this study is to understand the relationship between sleep disturbance and long-term mental health and functional recovery, as a step to improving the care, treatment and outcomes that people with TBI experience.

Primary Objective • To investigate the relationships between sleep disturbance, mental health outcomes and functional recovery in people with TBI.

Secondary Objectives

• To summarise what the literature indicates about how sleep disturbance impacts outcomes in recovery from TBI, including in the context of engagement with rehabilitation.

Part 1 - Cohort study

* To investigate the relationships between sleep disturbance and functional recovery at 3- and 6-months post-injury in people with TBI.
* To investigate the relationships between sleep disturbance and mental health at 3- and 6-months post-injury in people with TBI.
* To understand the impact of injury severity on mental health, and functional outcomes, in the context of sleep disturbance.
* To understand the fundamental properties of sleep disturbance for people who have sustained a TBI in the acute stage.

Part 2 - Cross-sectional study

* To investigate the relationships between chronic sleep disturbance, mental health and functional outcomes at over 1-year post-TBI.
* To understand how sleep disturbance and traumatic brain injury may impact on engagement with rehabilitation.
* To understand the fundamental properties of sleep disturbance for people who have sustained a TBI in the chronic stage.

Part 3 - Interviews

* To understand the human experience of TBI recovery and sleep disturbance.
* To explore people's perceptions of recovery and rehabilitation, in the context of TBI and sleep disturbance.

STUDY CONFIGURATION

This is a single-centre study taking place at Nottingham University Hospitals Trust (NUH). The configuration will be as follows:

Part 1

Cohort study with recruitment of those that meet the eligibility criteria from the Emergency Department and inpatient wards at NUH.

Part 2

Cross-sectional study design of those that meet the eligibility criteria recruited from Nottingham TBI community and outpatient rehabilitation teams at NUH.

Part 3

Semi-structured qualitative interviews using a sub-sample of participants from Part 1 and 2 studies.

DURATION OF THE STUDY AND PARTICIPANT INVOLVEMENT

Part 1 The recruitment process will begin once all approvals are in place, estimated to begin in September 2025 and end in February 2026. The follow-up time period will be 6 months for each participant, therefore, the estimated duration per participant will be 7 months. The total estimated study time is 12 months (completion in September 2026).

Participant involvement:

GENEActiv Device to be worn for a continuous 2 week period. Sleep diaries to be completed whilst participants are wearing the device, this will take approximately 5 minutes each day.

Questionnaires will take participants approximately 60 minutes to complete at the 3 and 6-month time points.

Part 2 The recruitment process is estimated to begin in March 2026, with a duration of 3 months. As data will be taken at a single time-point, the total duration of the study is estimated to be 4 months (completion in June 2026).

Participant involvement:

GENEActiv Device to be worn for a continuous 2 week period. Sleep diaries to be completed whilst participants are wearing the device, this will take approximately 5 minutes each day.

Questionnaires will take participants approximately 60 minutes to complete a single time point.

Part 3 Recruitment will take place by sampling from the 2 previous studies, with a planned start date of July 2026. Interviews will take place over 4-6 weeks, therefore the total study duration is estimated to be 6 weeks (completion in August 2026).

Participant involvement:

The interviews are estimated to take between 45-60minutes.

Recruitment

Participants will be recruited from one of the following departments at Nottingham University Hospitals Trust (NUH):

* The Emergency Department
* Neurosciences
* Major Trauma
* the National Rehabilitation Centre/ Linden Lodge Inpatient Rehab
* Nottingham TBI Team
* Nottingham Neuro Outpatient Services

The initial approach will be from a member of the patient's usual care team (which may include the investigator or research nurses at NUH). Participants will either be approached whilst they remain an inpatient at the hospital or post-discharge by their usual care team, by reviewing admissions by database and contacting participants by telephone, letter or email to gain consent to participate and determine study eligibility.

A sampling strategy will be in place to recruit participants across TBI severity, and to ensure diversity of the sample, such as across age and sex.

The investigator or their nominee, e.g. from the research team or a member of the participant's usual care team, will inform the participant of all aspects pertaining to participation in the study.

Participants will be given a chance to take the study information home if needed for further consideration or family consultancy. Participants will be excluded from the study anytime if they are unwilling to participate or unable to give informed consent.

If needed, the usual hospital interpreter and translator services will be available to assist with discussion of the study, the participant information sheets, and consent forms, but the consent forms and information sheets will not be available in other languages.

It will be explained to the potential participant that entry into the study is entirely voluntary and that their treatment and care will not be affected by their decision. It will also be explained that they can withdraw at any time but attempts will be made to avoid this occurrence. In the event of their withdrawal, it will be explained that their data collected so far cannot be erased and investigators will seek consent to use the data in the final analyses where appropriate.

STUDY REGIMEN

As this study is not a trial, there will be no individual treatments. All participants will wear the device for the specified time period and all participants will complete all outcome measures.

Part 1

Cohort study with recruitment of those that meet the eligibility criteria from the Emergency Department and inpatient wards at NUH:

* Participants will wear the GENEActiv activity tracker for a 2-week period, within 12 weeks of injury
* A sleep diary will be completed whilst participants are wearing the activity tracker. This will take approximately 5 minutes to complete each morning.
* Participants will send the GENEActiv device and the sleep diary back to study headquarters by signed and tracked, pre-paid post. There will also be the option of completing the sleep diary online via RedCap.
* Participants will complete questionnaire outcome measures, which will take approximately 60 minutes in total. This will be completed at 3 and 6-month time-points. Options will be to complete questionnaires over the telephone, online via RedCap or paper-based.
* A sample of participants will be asked to wear the activity tracker and complete sleep diaries for an additional 2 weeks as above, at the 6-month time point.

Part 2

Cross-sectional study design of those that meet the eligibility criteria recruited from Nottingham TBI community and outpatient rehabilitation teams at NUH. Participants must have sustained their injury more than 12 months ago.

* Participants will wear the GENEActiv activity tracker for a 2-week period.
* A sleep diary will be completed whilst participants are wearing the activity tracker. This will take approximately 5 minutes to complete each morning.
* Participants will send the GENEActiv device and the sleep diary back to study headquarters by signed and tracked, pre-paid post. There will also be the option of completing the sleep diary online via RedCap.
* Participants will undertake questionnaire outcomes measures at a single time point. This will take approximately 60 minutes in total. Options will be to complete questionnaires over the telephone, online via RedCap or paper-based.
* Clinicians will be recruited via their line manager via letter or email, and will be staff that have been working with participants within rehabilitation services. They will complete questionnaires to explore the individual's engagement with rehabilitation. The questionnaire will take clinicians approximately 2-3 minutes to complete per participant and can be completed online, over the telephone or paper-based.

Part 3

Semi-structured interviews will take place with a sample of the participants with TBI from Parts 1 and 2. Interviews will be conducted by Research Co-Investigator Irene Morgan-Brown, who is a clinician experienced in working with people with brain injuries. They will be conducted either online, in-person or over the telephone, at the preference of the participant. Interviews are estimated to take 45-60 minutes per participant. Interviews may involve sensitive topics, and there will be a distress management plan in place to help signpost participants, if needed. Breaks will also be offered to participants during the interview. Interviews will be recorded with an audio recording device. Once interviews have taken place, data recordings will be uploaded to the secure study database. Any data associated with interviews will be treated as source data and will be retained in study archives, with personal identifiers removed.

Further information regarding the GENEActiv device:

Participants will be provided with the device once they have consented to take part in the study. The device will either be given to them by the research team whilst they remain an inpatient in hospital, or the device will be sent to them via signed and tracked post. The participants will be asked to wear the device at all times, and it will record sleep and movement via actigraphy. The device is fully waterproof. Once participants have worn the device for the 2-week period, they will send it back to study headquarters via signed and tracked pre-paid post. Raw data from the device will then be downloaded onto a secure server with GENEActiv software by the research team. No personal identifiers or location data will be used or recorded on the software.

STATISTICS

Methods

The Co-Investigator Irene Morgan-Brown will evaluate the findings using Jamovi software. Support will be sought from the Chief Investigator and Co-Investigators as appropriate. Statistics guidance from a statistician will also be sought from the School of Health Sciences Statistics Drop-In sessions. The analysis will take place on the University of Nottingham computer and backed up on University of Nottingham servers.

Initially, correlation analysis will be conducted to determine the strongest relationships between sleep variables and each functional or mental health outcome. Then, multivariate regression analysis methods will be applied to control for confounders and explore the predictive quality of sleep disturbance on outcomes. Injury severity will also be included in the model to determine whether it impacts the relationship between the sleep predictors and the outcome measures.

Qualitative data will be analysed using thematic analysis, which will involve identifying themes across all transcripts.

A sequential explanatory mixed methods approach will be used. Each phase of the research will be analysed individually and then inform the next stage. For example, the interview guide will be developed based on the results of the quantitative study. Data across all study elements will be integrated through a narrative convergence matrix.

Sample size and justification

Previous research that is directly relevant to our question with a TBI cohort is not available. As such, we have powered the study based on identified links between sleep and mental health measures in other clinical cohorts. Rao et al. (2008) indicated an effect size of 0.13 when exploring the relationship between sleep disturbance and mental health outcome (Rao et al. 2008). Similarly, Fleming et al. (2021) and Rao et al. (2020) found effect sizes of 0.19 and 0.32 when linking sleep with depression and anxiety, respectively.

Taking a medium effect size (0.15) in accordance with these studies, 6 predictor variables (age, sex, TBI severity and 3 sleep measures identified as described below), a sample size of 43 participants is needed (G*Power 3.1.9.7, Linear Multiple Regression, α = 0.05, 80% power). Accounting for an expected drop-out rate of 20%, investigators would need to aim to recruit 54 participants.

However, in general approximately 10 participants per predictor variable are suggested for linear regression analyses. Investigators will therefore round up and aim for a minimum recruitment of 60 participants to each study.

For Part 1, investigators will aim to recruit 120 participants, due to the high volume of head injuries admitted to the Emergency Department and the wider range of injury severity. For Part 2, investigators will aim to recruit 60 participants. Therefore, a total of 180 participants will be recruited for the study.

Feature selection: Investigators will acquire a broad set of sleep measures including subjective (questionnaires) and objective (actigraphy) metrics. In order to identify the most relevant of these variables, and to keep the overall number of predictors low for the linear regression analysis, we will perform correlation analyses between the sleep variables and the outcome measures. The 3 most highly correlated predictors for each outcome will be retained for the linear regression analysis.

Part 3

For interviews, study size estimate is based on conducting in-depth semi-structured interviews and theoretical underpinning of information power. Therefore, a sample size of approximately 15-20 participants is estimated.

USER AND PUBLIC INVOLVEMENT

Public and Patient Involvement (PPI) has taken place and been fundamental in refining and developing the study design, to ensure that the study is appropriate and relevant to those who have lived experience of TBI.

There is an active PPI Group of individuals with lived experience of TBI that have been consulted in the development of the design and protocol, and will continue to be consulted throughout the research process. For example, they have fed back their opinions on what outcomes are important to focus on for this study. PPI group members have also reviewed relevant documents, such as the participant information sheets, to ensure they are appropriate for the patient group.

STUDY FINANCES

Funding source This study is funded by the Wellcome Trust as part of the Midlands Mental Health and Neurosciences Doctoral Training Programme.

Participant stipends and payments Participants will not be paid to participate in the study. Travel expenses will be offered for any hospital visits in excess of usual care.

ELIGIBILITY:
Part 1

Inclusion criteria:

* Age 18-60 years
* Patients presenting to the Emergency Department within 24 hours of head injury
* Medically diagnosed TBI of any severity
* Glasgow Coma Scale (GCS) score documented on admission
* Able to provide informed consent to take part in the study
* To be able to wear an activity tracker for a period of 2 weeks, in usual home environment within 12 weeks of injury

Exclusion criteria:

* Unable to understand the study requirements or give informed consent
* Other diagnosed neurological condition such as, but not limited to, stroke, brain tumour, epilepsy, motor neuron disease, Parkinson's disease, or spinal cord injury
* No definition of TBI or description of TBI severity, patient report only, or unknown time since injury
* Pre-existing sleep disorder (self-reported or from clinical records)
* Individuals that have working patterns that include night shifts
* Not contactable via telephone, letter or email

Part 2

Inclusion criteria:

* Age 18-60 years
* Medically diagnosed TBI of any severity
* Glasgow Coma Scale (GCS) score documented in medical notes
* Able to provide informed consent to take part in the study
* TBI sustained >12 months
* Able to wear an activity tracker in usual home environment for a period of 2 weeks

Exclusion criteria:

* Unable to understand the study requirements or give informed consent
* Other diagnosed neurological condition such as, but not limited to, stroke, brain tumour, epilepsy, motor neuron disease, Parkinson's disease, or spinal cord injury
* No definition of TBI or description of TBI severity, patient report only, or unknown time since injury
* Pre-existing sleep disorder (self-reported or from clinical records)
* Individuals that have working patterns that include night shifts
* Not contactable via telephone, letter or email

Part 2 - For clinicians

Inclusion criteria:

* A registered healthcare professional working at Nottingham University Hospitals Trust
* Clinical experience of delivering rehabilitation services to participants with TBI that have been recruited to the study

Exclusion criteria:

* Not contactable via telephone, letter or email
* Unable to understand the study requirements or give informed consent

Part 3

• Inclusion/Exclusion criteria as stated above. 50% of participants will be recruited from Part 1, and 50% of participants will be recruited from Part 2 for both studies.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: People with traumatic brain injury, recruited from the following locations:
  Nottingham University Hospitals Trust, to include:
  * Emergency Department (Queens Medical Centre)
  * Neurosciences and Major Trauma wards (Queens Medical Centre)
  * Linden Lodge Inpatient Neuro Rehab / National Rehabilitation Centre (City Hospital and Stanford Hall)
  * Nottingham TBI Community Rehabilitation Team (City Hospital)
  * Nottingham Neuro Rehabilitation Outpatient team (City Hospital)
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Functional outcome | Part 1: 3 and 6 months post-injury Part 2: At any point between Day 1 - 28
  Standardised and validated questionnaire: Extended Glasgow Outcome Score (GOSE)
Functional outcome | Part 1: 3 and 6 months post-injury Part 2: At any point between Day 1-28
  Standardised and validated questionnaire: Quality of Life after Brain injury (QOLIBRI)

SECONDARY OUTCOMES:
Mental health outcome | Part 1: 3 and 6 months post-injury For Part 2: At any point between Day 1-28
  Standardised and validated questionnaire: Patient Health Questionnaire (PHQ-9)
Mental health outcome | Part 1: 3 and 6 months post-injury For Part 2: At any point between Day 1-28
  Standardised and validated questionnaire: General Anxiety Disorder-7 (GAD-7)
Mental health outcome | Part 1: 3 and 6 months post-injury For Part 2: At any point between Day 1-28
  Standardised and validated questionnaire: Post Traumatic Stress Disorder Checklist 5 (PCL-5)
Rehabilitation engagement outcome | For Part 2: At any point between Day 1-28
  Standardised and validated questionnaire: Hopkins Rehabilitation Engagement Rating Scale (HRERS). Completed by clinicians working with participants recruited into the study.
Subjective sleep disturbance outcome | Part 1: 3 and 6 months post-injury For Part 2: At any point between Day 1-28
  Standardised and validated questionnaire: Pittsburgh Sleep Quality Index (PSQI)

OTHER OUTCOMES:
Exposure of interest | For Part 1: Within 12 weeks of injury, for a 2 week period For Part 2: At over 12 months of injury, for a 2 week period
  Actigraphy of sleep data from the GENEActiv device:
  • Total Sleep Duration (mm:hh)
Exposure of interest | For Part 1: Within 12 weeks of injury, for a 2 week period For Part 2: At over 12 months of injury, for a 2 week period
  Actigraphy of sleep data from the GENEActiv device:
  • WASO (Wake After Sleep Onset) (mm:hh)
Exposure of interest | For Part 1: Within 12 weeks of injury, for a 2 week period For Part 2: At over 12 months of injury, for a 2 week period
  Actigraphy of sleep data from the GENEActiv device, including:
  • Sleep Efficiency (%)
Exposure of interest | For Part 1: Within 12 weeks of injury, for a 2 week period For Part 2: At over 12 months of injury, for a 2 week period
  Actigraphy of sleep data from the GENEActiv device:
  • Sleep Onset Latency (hh:mm)

CONTACTS AND LOCATIONS:
Overall Officials: Professor Holly Blake, Study Chair — University of Nottingham; Professor Andrew Bagshaw, Study Director — University of Birmingham; Dr Karen Mullinger, Study Director — University of Nottingham
Locations (1):
- Nottingham University Hosptials Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided